CLINICAL TRIAL: NCT02030301
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation, Phase 1/2 Trial to Evaluate the Safety and Efficacy of Herpes Simplex Virus, Type 2 Therapeutic DNA Vaccines in Symptomatic HSV-2-Seropositive Adults
Brief Title: Safety and Efficacy Trial of DNA Vaccines to Treat Genital Herpes in Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSV2-101
Record Dates: First submitted 2013-12-20; First posted 2014-01-08 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Genital Herpes Simplex Type 2
Keywords: Herpes Simplex Virus, Type 2; Herpes; HSV-2
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- VCL-HB01, 0.25-mL dose (Experimental): VCL-HB01, 0.25-mL dose by intramuscular injection once every 28 days for 3 doses
  Interventions: Biological: VCL-HB01
- PBS, 0.25-mL dose (Placebo Comparator): PBS, 0.25-mL dose by intramuscular injection once every 28 days for 3 doses
  Interventions: Biological: PBS
- VCL-HB01, 0.5-mL dose (Experimental): VCL-HB01, 0.5-mL dose by intramuscular injection once every 28 days for 3 doses
  Interventions: Biological: VCL-HB01
- PBS, 0.5-mL dose (Placebo Comparator): PBS, 0.5-mL dose by intramuscular injection once every 28 days for 3 doses
  Interventions: Biological: PBS
- VCL-HB01, 1-mL dose (Experimental): VCL-HB01, 1-mL dose by intramuscular injection once every 28 days for 3 doses
  Interventions: Biological: VCL-HB01
- VCL-HM01, 1-mL dose (Experimental): VCL-HM01, 1-mL dose by intramuscular injection once every 28 days for 3 doses
  Interventions: Biological: VCL-HM01
- PBS, 1-mL dose (Placebo Comparator): PBS, 1-mL dose by intramuscular injection once every 28 days for 3 doses
  Interventions: Biological: PBS

INTERVENTIONS:
Biological: VCL-HB01 — Plasmid DNA vaccine encoding two HSV-2 proteins; formulated with Vaxfectin®
  Arms: VCL-HB01, 0.25-mL dose; VCL-HB01, 0.5-mL dose; VCL-HB01, 1-mL dose
Biological: VCL-HM01 — Plasmid DNA vaccine encoding one HSV-2 protein; formulated with Vaxfectin®
  Arms: VCL-HM01, 1-mL dose
Biological: PBS — Phosphate-buffered saline
  Arms: PBS, 0.25-mL dose; PBS, 0.5-mL dose; PBS, 1-mL dose

SUMMARY:
The purpose of this study is to test the safety and effectiveness of two experimental therapeutic vaccines against herpes simplex virus, type 2 (HSV-2).

DETAILED DESCRIPTION:
This is a dose escalation study to evaluate the safety, immunogenicity, and efficacy of 3 doses of HSV plasmid DNA (pDNA) vaccines formulated with Vaxfectin® in subjects with a minimum of 1 year of reported history of genital herpes, and either 2 to 9 recurrences within the year prior to screening, or 2 to 9 recurrences per year prior to starting suppressive therapy.

ELIGIBILITY:
Inclusion Criteria:

* HSV-2 seropositive
* A minimum of 1 year of reported history of genital herpes and either 2 to 9 recurrences within the year prior to screening or 2 to 9 recurrences per year prior to starting suppressive therapy

Exclusion Criteria:

* History of receiving an investigational HSV vaccine
* Chronic illness for which a subject's immune system is suspected to be impaired or altered, such as cancer, autoimmune conditions, or diabetes
* Pregnant or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to Day 420
Viral shedding rate change from baseline | Baseline, Day 150

SECONDARY OUTCOMES:
Genital lesion rate change from baseline | Baseline, Day 150
HSV DNA copy numbers change from baseline | Baseline, Day 150
Genital recurrence rate compared with placebo | Up to Day 330
Subclinical genital shedding rate change from baseline | Up to Day 150
T-cell and/or antibody responses change from baseline | Baseline, Days 7, 35, 63, 150, 330

OTHER OUTCOMES:
Genital shedding rate change from baseline over time | Baseline, Day 330
Genital lesion rate change from baseline | Baseline, Day 330
Subclinical genital shedding rate change from baseline | Baseline, Day 330

CONTACTS AND LOCATIONS:
Overall Officials: Mammen P. Mammen, Jr., MD, FIDSA, Study Director — Vical
Locations (7):
- United States (7):
  - Alabama Vaccine Research Clinic, Birmingham, Alabama
  - Broward Research Group, Hollywood, Florida
  - Indiana University Infectious Diseases Research, Indianapolis, Indiana
  - Westover Heights Clinic, Portland, Oregon
  - Center for Clinical Studies, Houston, Texas
  - University of Utah - Division of Infectious Diseases, Salt Lake City, Utah
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No